CLINICAL TRIAL: NCT00890201
Title: Is Pancreaticobiliary Reflux in Patients With Cholelithiasis and Without Cholelithiasis a Normal Phenomenon?
Brief Title: Pancreaticobiliary Reflux in Patients Without Cholelithiasis
Status: Completed | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: MARCELO A. BELTRAN, M.D., HOSPITAL DE LA SERENA
Other Study IDs: HLS-2704009-02
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Results first posted 2009-10-20 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-09

CONDITIONS: Pancreaticobiliary Reflux
Keywords: Pancreaticobiliary reflux; Normal pancreaticobiliary junction; Gallstones; Cholelithiasis; Cholecystectomy
MeSH Terms: conditions — Gallstones; Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Gallbladder: Patients with normal gallbladder (without gallstones) evidenced by preoperative ultrasonography (and postoperative biopsy) submitted to elective gastroesophageal surgery (gastrectomy for gastric cancer, bariatric surgery or esophageal surgery such as Nissen plicature or miotomy for achalasia).
  The pancreaticobiliary junction must be normal as evidenced by intraoperative cholangiography. Preoperative values of amylase and lipase must be normal.
  Interventions: Procedure: Gallbladder bile sampling and intraoperative cholangiography
- Gallbladder with gallstones: Patients submitted to elective cholecystectomy for diseased gallbladders (gallbladder with gallstones evidenced by preoperative ultrasound).
  The pancreaticobiliary junction must be normal as evidenced by intraoperative cholangiography and the preoperative amylase and lipase levels must also be normal.
  Interventions: Procedure: Gallbladder bile sampling and intraoperative cholangiography

INTERVENTIONS:
Procedure: Gallbladder bile sampling and intraoperative cholangiography — Interventions were exactly similar for both groups, and that is how it was intended to be:
  Gallbladder bile sampling: Sample 5 cc of gallbladder bile after the cystic duct has been clipped or ligated.
  Intraoperative cholangiography: Perform cholangiography before the cholecystectomy is finished
  Other Names: Measurement of pancreaticobiliary reflux

SUMMARY:
Pancreaticobiliary reflux has been found in patients with cholelithiasis and gallbladder cancer associated with normal pancreaticobiliary union. However, the presence of pancreaticobiliary reflux has not been studied in patients without gallstones (healthy gallbladders).

The authors believe that pancreaticobiliary reflux might be a normal phenomenon in patients with and without gallstones, although in patients with cholelithiasis it might constitute a pathological condition associated with dismotility of the biliary tree and the sphincter of Oddi.

DETAILED DESCRIPTION:
The objective of this study is to measure the levels of amylase and lipase in gallbladder bile of patients without gallstones and compare these values to the values of amylase and lipase of patients with gallstones and normal pancreaticobiliary union evidenced by intraoperative cholangiography.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 15 years of age
* Elective surgery
* Normal intraoperative cholangiography
* Normal preoperative serum amylase and lipase values

Exclusion Criteria:

* Common bile duct stones
* Anatomic anomalies at the pancreaticobiliary junction evidenced by intraoperative cholangiography
* Altered preoperative amylase and lipase levels
* Altered preoperative hepatic function tests
* Emergency surgery

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients with gallstones (symptomatic cholelithiasis) submitted to elective surgery.
  2. Patients without gallstones submitted to elective surgery for benign or malignant gastroesophageal diseases
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MARCELO A BELTRAN, M.D., Principal Investigator — Hospital de La Serena
Locations (1):
- Hospital de La Serena, La Serena, Coquimbo Region, Chile

REFERENCES:
- [Background] Beltran MA, Vracko J, Cumsille MA, Cruces KS, Almonacid J, Danilova T. Occult pancreaticobiliary reflux in gallbladder cancer and benign gallbladder diseases. J Surg Oncol. 2007 Jul 1;96(1):26-31. doi: 10.1002/jso.20756. PMID 17345616
- [Derived] Beltran MA, Contreras MA, Cruces KS. Pancreaticobiliary reflux in patients with and without cholelithiasis: is it a normal phenomenon? World J Surg. 2010 Dec;34(12):2915-21. doi: 10.1007/s00268-010-0771-2. PMID 20811747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at the Department of Surgery of the Hospital de La Serena from January 2009 to July 2009
Pre-assignment Details: Patients submitted to elective cholecystectomy for symptomatic gallstone disease, older than 16 years of age and patients submitted to elective gastrectomy for gastric cancer harboring normal gallbladders (without gallstones), were included in this trial. Patients within any other clinical situation were excluded
Period: Overall Study
Arm/Group | Normal Gallbladder | Gallbladder With Gallstones
Started | 38 (5 patients with gastric cancer and gallstone disease) | 159 (41 patients with acute cholecystitis and 15 patients with common bile duct stones)
Completed | 33 (33 patients with gastric cancer and without gallstone disease) | 103 (103 patients without acute cholecystitis or common bile duct stones)
Not Completed | 5 | 56
Not completed — Protocol Violation | 5 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Gallbladder | Gallbladder With Gallstones | Total
Number analyzed (Participants) | 38 | 159 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 33 | 149 | 182
  >=65 years | 5 | 8 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10) | 43.4 (12.6) | 46.3 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 17 | 140 | 157
Region of Enrollment [Number; unit: participants]
  Chile | 38 | 159 | 197

OUTCOME MEASURES:

1. Primary Outcome: Amylase and Lipase Values in Gallbladder Bile
Description: Normal values of lipase and amylase in gallbladder bile should be zero
Time Frame: 24 hours
Population: The number of participants analyzed was determined by the number of participants that matched the inclusion criteria. As posted elsewhere some participants were excluded from this analysis based in the exclusion criteria of the protocol.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Normal Gallbladder | Gallbladder With Gallstones
Number analyzed (Participants) | 33 | 103
mg/dl
  Amylase | 5.5 (16.4) | 181.2 (352)
  Lipase | 9.5 (16.6) | 434.8 (1224)

2. Secondary Outcome: Amylase and Lipase Values in Normal Gallbladders
Time Frame: 24 hours
Reporting Status: Not Posted

3. Secondary Outcome: Amylase and Lipase Values in Gallbladders With Cholelithiasis
Time Frame: 24 hours
Reporting Status: Not Posted

4. Secondary Outcome: Normal Operative Cholangiography
Time Frame: 24 hours
Reporting Status: Not Posted

5. Secondary Outcome: Normal Preoperative Serum Values of Amylase and Lipase
Time Frame: 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse events were not assessed
Arm/Group | Normal Gallbladder | Gallbladder With Gallstones
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes